CLINICAL TRIAL: NCT06151808
Title: An Open-label, Non-randomized, Single-center Study, Evaluating the Imaging Characteristics of XTR006 Injection in Non-cognitively Impaired Subjects, MCI Due to Alzheimer Disease (AD), and Mild to Moderate AD Subjects
Brief Title: Analysis of XTR006 PET Imaging in Non-cognitively Impaired Subjects, MCI Due toAD, and Mild to Moderate AD Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinotau Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STB-XTR006-IIT-01
Record Dates: First submitted 2023-08-25; First posted 2023-11-30 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Alzheimer Disease
Keywords: Tau PET; Dosimetry; Alzheimer's disease; Chinese; XTR006
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: 30 subjects with non-cognitive impairment, 30 subjects with MCI due to AD， 30 subjects with mild to moderate AD.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- non-cognitive impairment (Sham Comparator): 30 subjects with non-cognitive impairment
  Interventions: Drug: XTR006
- AD-derived MCI (Experimental): 30 subjects with AD-derived MCI
  Interventions: Drug: XTR006
- mild to moderate AD. (Experimental): 30 subjects with mild to moderate AD.
  Interventions: Drug: XTR006

INTERVENTIONS:
Drug: XTR006 — All participants will receive a single intravenous dose of 8.0-10.0mCi of XTR006 followed by PET scan

SUMMARY:
This is an investigator-initiated clinical (IIT)study.The main purpose of this study was to evaluate the diagnostic efficacy of XTR006 PET qualitative reading and quantitative analysis in detecting mild cognitive impairment（MCI）due to AD and mild to moderate AD based on clinical diagnosis, and to establish XTR006 PET imaging parameters and qualitative reading and quantitative analysis methods.

DETAILED DESCRIPTION:
XTR006 is a 18F-labeled PET tracer, for the quantification of neurofibrillary tangle (NFT) deposition in the brain. Brain NFT deposition is a pathologic finding in Alzheimer's Disease (AD), with brain NFT density shown to correlate with the severity of cognitive impairment in AD. 90 Chinese subjects (30 subjects with non-cognitive impairment, 30 subjects with MCI due to AD and 30 subjects with mild to moderate AD) who meet all of the inclusion and none of the exclusion criteriawill be enrolled in this IIT study. Subjects will receive 8-10mCi of XTR006 via IV injection. qualitative reading and quantitative analysis methods will be investigated. Safety and tolerability will be observed.

ELIGIBILITY:
Inclusion Criteria:

* 1. Inclusion criteria for non-cognitively impaired subjects

  1. Male or female aged between 55 to 85 years old (including 50 and 85 years old);
  2. Clinical dementia score (CDR) of 0;
  3. the Mini-Mental State Examination Scale (MMSE score) of ≥28;
  4. Aβ PET imaging is negative;
  5. Able to cooperate with the tests required for research including neuropsychological tests (cognitive ability, language ability, visual and auditory acuity can meet the requirements of the test);
  6. The researcher judges that the subjects are in good health, and there is no abnormal or abnormality in the comprehensive physical examination, vital sign examination and laboratory examination, but they can participate in this bridging clinical trial according to the judgment of the clinician;
  7. For women of potential fertility (not yet or within 2 years of menopause), effective contraceptive measures must be used during the study period and within 6 months after the end of the study (effective contraceptive measures refer to sterilization, intrauterine hormonal devices, contraception condoms, contraceptives/dose, abstinence or partner removal of the vas deferens, etc.); male subjects should agree to use contraceptives during the study period and within 6 months after the end of the study period;
  8. Able to sign the informed consent form.
* 2. Inclusion criteria for MCI due to AD

  1. Male or female aged between 55-85 years old (including 50 and 85 years old);
  2. Diagnosed as MCI due to AD according to NIA-AA standard in 2011;
  3. Have symptoms of subjective memory loss and maintain independent ability of daily life;
  4. MMSE score≤27;
  5. CDR score=0.5;
  6. Aβ PET imaging is positive;
  7. Able to cooperate with the tests required for research including neuropsychological tests (cognitive ability, language ability, visual and auditory acuity can meet the requirements of the test);
  8. For women of potential fertility (not yet or within 2 years of menopause), effective contraceptive measures must be used during the study period and within 6 months after the end of the study (effective contraceptive measures refer to sterilization, intrauterine hormonal devices, contraception condoms, contraceptives/dose, abstinence or partner removal of the vas deferens, etc.); male subjects should agree to use contraceptives during the study period and within 6 months after the end of the study period;
  9. Able to sign the informed consent form.
* 3. Inclusion criteria for subjects with mild to moderate AD

  1. Male or female aged between 50-85 years old (including 55 and 85 years old);
  2. Diagnosed as probable AD according to NIA-AA standard in 2011;
  3. MMSE score≤27
  4. 1≤CDR score≤2;
  5. Aβ PET imaging is positive;
  6. Have the ability to complete the cognitive ability test and other tests specified in the protocal;
  7. The investigator judges that the subject's "caregiver" can provide accurate information and report on the patient's cognitive and functional abilities;
  8. For women of potential fertility (not yet menopause or within 2 years of menopause), effective contraceptive measures must be used during the study period and within 6 months after the end of the study (effective contraceptive measures refer to sterilization, intrauterine hormonal devices, contraception condoms, contraceptives/dose, abstinence or partner removal of the vas deferens, etc.); male subjects should agree to use contraceptives during the study period and within 6 months after the end of the study period;
  9. Able to sign the informed consent form.

Exclusion Criteria:

* 1. Exclusion criteria for non-cognitively impaired subjects

  1. years of education ≤6 years;
  2. Severe neurological diseases, such as cerebrovascular diseases, inflammatory or infectious diseases, or any metabolic encephalopathy, neurodegenerative diseases, including Parkinson's disease history or physical or imaging manifestations;
  3. History of severe craniocerebral injury, craniocerebral surgery or intracranial hematoma with permanent brain injury;
  4. The results of cranial magnetic resonance imaging (MRI) also meet the following imaging findings: ①There are two or more infarcts outside the brain stem (diameter greater than 2 cm); ②Key parts such as thalamus, hippocampus, entorhinal cortex and angular gyrus Lacunar infarction; ③Fazekas score of high white matter damage ≥4;
  5. Brain MRI examination showed enlarged perivascular space with subcortical diameter >3mm in short axis;
  6. SWI (susceptibility-weighted imaging) prompts: cerebral microbleeds ≥8 locations;
  7. History of alcohol or drug abuse/dependence;
  8. Contraindications of MRI examination: such as heart pacemaker or nerve stimulator or metal foreign body, high fever, etc.;
  9. Invasive surgery is planned within one week after administration of the study drug;
  10. Allergy to the investigational drug or any of its components and/or a history of severe allergic reaction to the drug or allergens (such as history of alcohol allergy or allergic asthma);
  11. Any major disease or unstable disease state (such as unstable angina pectoris, myocardial infarction or coronary revascularization, heart failure, acute and chronic renal failure, chronic liver disease, severe lung disease, blood disease, poor blood sugar control, chronic infection in the past 2 years, received surgical treatment 7 days ago, advanced cardiac insufficiency (New York Heart Association (NYHA stage IV), etc.);
  12. History of tumor within 5 years (except cervical carcinoma in situ, prostate carcinoma in situ or local skin cancer after surgery);
  13. Human immunodeficiency virus (HIV), hepatitis C or Treponema pallidum antibody test positive, hepatitis B surface antigen positive (except hepatitis B carriers);
  14. Received drug therapy or other treatments (such as chemotherapy) that cause large fluctuations in hematological or biochemical indicators or serious side effects within two weeks before the screening examination;
  15. Receive any contrast agent or radiopharmaceutical within 48 hours before application of test drug, or will use contrast agent within 24 hours after administration of study drug;
  16. Participated in clinical research of other drugs within 30 days before enrollment or within 5 half-lives of the study drug (whichever is longer), and/or used any radiopharmaceuticals before the administration of the study drug, and not more than 10 radioactive half-lives apart;
  17. History of epilepsy;
  18. History of electroconvulsive therapy;
  19. History of delirium (e.g. after surgery);
  20. Other investigators deem it inappropriate to participate in the trial.
* 2. Exclusion criteria for subjects with MCI due to AD and mild to moderate AD

  1. years of education ≤6 years;
  2. Epilepsy episode occurred within the past 1 year;
  3. Dementia caused by other reasons or cognitive dysfunction caused by other reasons: such as vascular dementia, Parkinson's disease dementia, Lewy body dementia, normal intracranial pressure hydrocephalus, intracranial mass, central nervous system infection (Such as HIV, syphilis, etc.), metabolic encephalopathy, etc.;
  4. The results of cranial MRI also meet the following imaging findings: ①There are more than two infarcts outside the brain stem (diameter greater than 2 cm); ②Lacunar infarction in key parts such as the thalamus, hippocampus, entorhinal cortex and angular gyrus ③The Fazekas score of high white matter damage ≥ 4;
  5. Brain MRI examination showed enlarged perivascular space with subcortical diameter >3mm in short axis;
  6. SWI prompt: cerebral microbleeds ≥8 locations;
  7. History of alcohol or drug abuse/dependence;
  8. Contraindications of MRI examination: such as heart pacemaker or nerve stimulator or metal foreign body, high fever, etc.;
  9. Subjects who plan to undergo surgery and/or other invasive surgery within 24 hours after the application of the trial drug;
  10. Allergy to the investigational drug or any of its components and/or history of severe allergic reaction to the drug or allergens (such as history of alcohol allergy or allergic asthma);
  11. Any major disease or unstable disease state (such as unstable angina pectoris, myocardial infarction or coronary revascularization, heart failure, acute and chronic renal failure, chronic liver disease, severe lung disease, blood Diabetic patients with disease, poor blood sugar control, chronic infection in the past 2 years, received surgical treatment 7 days ago, advanced cardiac insufficiency (NYHA stage IV), major depressive episode, etc.);
  12. History of tumor within 5 years (except cervical carcinoma in situ, prostate carcinoma in situ or local skin cancer after surgery);
  13. HIV, hepatitis C or Treponema pallidum antibody test positive, hepatitis B surface antigen positive (except hepatitis B carriers);
  14. History of severe craniocerebral injury, craniocerebral surgery or intracranial hematoma with permanent brain injury;
  15. Received drug therapy or other treatments (such as chemotherapy) that cause large fluctuations in hematological or biochemical indicators or serious side effects within two weeks before the screening examination;
  16. Receive any contrast agent or radiopharmaceutical within 48 hours before application of test drug, or will use contrast agent within 24 hours after administration of test drug;
  17. Participated in clinical research of other drugs within 30 days before enrollment or within 5 half-lives of the study drug (whichever is longer), and/or used any radiopharmaceuticals before the administration of the study drug, and not more than 10 radioactive half-lives apart;
  18. Other investigators deem it inappropriate to participate in the trial.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
To investigate the sensitivity and specificity of XTR006 PET imaging by reading | day 1
  Sensitivity and specificity of XTR006 PET images for diagnosis of MCI and AD will be measured by comparison to the standard of truth (SoT) obtained through standard of care clinical diagnosis.
To investigate the sensitivity and specificity of XTR006 PET imaging by SUVR | day 1
  Sensitivity and specificity of XTR006 PET images for diagnosis of MCI and AD will be measured by comparison to the standard of truth (SoT) obtained through standard of care clinical diagnosis.

SECONDARY OUTCOMES:
To investigate the parameters of XTR006 PET imaging in the brain | 0 to 130 minutes post injection
  PET images were collected 0-130min after a single intravenous administration of XTR006, and the start time when the SUVR value of Braak brain region was stable with cerebellar gray matter as the reference area was analyzed
To investigate the methodology of XTR006 PET qualitative reading | day 1
  Sensitivity and specificity of different XTR006 PET qualitative reading rules for diagnosis of MCI and AD.
To investigate the consistency among XTR006 PET readers and the reproducibility of the readers themselves. | day 1
  Kappa value between XTR006 PET images readers and Kappa value of readers themselves.
To investigate the quantitative analysis methodology of XTR006 PET. | day 1
  SUVR cut off value and Sensitivity/specificity of different XTR006 PET quantitative analysis rules for diagnosis of MCI and AD.
Descripte study product-related adverse events by numbers,degree and kinds as assessed by CTCAE v5.0 | up to 7days
  Safety Observation: Number of participants with adverse events and severe adverse events after drug injection.

CONTACTS AND LOCATIONS:
Overall Officials: jianjun jia, Ph.D, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China